CLINICAL TRIAL: NCT01096628
Title: Chiropractic and Exercise for Low Back Pain in Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: University of Western States (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HP15124
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Low Back Pain
Keywords: adolescent; low back pain; chiropractic; exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chiropractic + Exercise (Experimental)
  Interventions: Other: Chiropractic + Exercise
- Exercise (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Chiropractic + Exercise — Treatment will include eight to 16 treatments provided over the 12-week period. Each treatment visit will last from 10-20 minutes and consist of manual spinal manipulation and mobilization. Light soft tissue techniques (i.e., active and passive muscle stretching, hot and cold packs, and ischemic compression of tender points) will be used as indicated to facilitate the manual therapy.
  Patients will attend 8 to 16, one-on-one, 45-minute sessions over the course of 3 months. The sessions will follow a standardized approach but will be individualized to meet the patient's needs specific to their lifestyle, fitness level, and clinical characteristics. The exercise program will be comprised of three parts: 1) education, 2) supervised exercise, and 3) home exercise.
  Arms: Chiropractic + Exercise
Other: Exercise — Patients will attend 8 to 16, one-on-one, 45-minute sessions over the course of 3 months. The sessions will follow a standardized approach but will be individualized to meet the patient's needs specific to their lifestyle, fitness level, and clinical characteristics. The exercise program will be comprised of three parts: 1) education, 2) supervised exercise, and 3) home exercise.
  Arms: Exercise

SUMMARY:
Recent research has confirmed that low back pain (LBP) is a significant health problem not only for adults, but also for children and adolescents. Given the enormous social and economic costs associated with LBP, it is critical that attempts be made to decrease the burden of LBP for patients and society.

The primary aim of this project is to determine the relative clinical effectiveness of 3 months of chiropractic care and supervised exercise versus supervised exercise in 184 adolescents with sub-acute recurrent, or chronic LBP. Relative effectiveness will be evaluated in the short, intermediate and long term using pain as the primary outcome measure. Secondary aims are to assess group differences in patient self-reported disability, quality of life, perceived improvement, satisfaction, activity levels, lumbar dynamic motion, and trunk muscle endurance. Patients' and caregivers' perceptions of treatment using qualitative interviews will also be assessed.

DETAILED DESCRIPTION:
This study is a two-site, prospective, parallel group, observer-blinded randomized controlled trial (RCT). The objective of this study is to determine the relative clinical effectiveness of 1) chiropractic care and supervised exercise; and 2) supervised exercise in adolescents with sub-acute recurrent LBP (2-12 weeks duration) or chronic LBP (>12 weeks duration ).

A total of 184 participants 12-18 years of age will be recruited from the Twin Cities of Minneapolis/St.Paul and Portland metropolitan areas to the research clinics at Northwestern Health Sciences University (NWHSU) and the University of Western States Portland(UWS). Data collection measures and study protocols will be standardized across sites. The Office of Data Management at NWHSU will serve as the central data coordinating center, with a web-based interface for centralized data handling and treatment assignment.

Self-reported outcome measures assessing pain and disability, will be collected at baseline, 1, 2, 3, 4, 5, 6, and 12 months post-randomization. In addition, quality of life, improvement, and satisfaction will be measured at months 3, 6 and 12. Objective outcome measures including lumbar dynamic motion and trunk muscle endurance will be assessed by blinded examiners at baseline and post-treatment phase (3 and 6 months). Patients will wear accelerometers for the 7 days preceding follow up visits for months 3 and 6. Qualitative patient interviews assessing patient and care-giver perceptions of care will be also be conducted at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age
* Stable prescription medication plan (no changes in prescription medications that affect musculoskeletal pain in the previous month)
* Primary complaint of low back pain > 3 on 0 to 10 scale

Either:

* Recurrent, sub-acute low back pain defined as current episode of 2-12 weeks duration AND at least an additional 10 days of back pain in the past year OR
* Chronic low back pain defined as current episode >12 weeks duration

Exclusion Criteria:

* Chiropractic care or exercise therapy in the previous month
* Ongoing treatment for low back pain by other health care providers
* Other serious physical or mental health care conditions (for example diabetes, cancer, etc.)
* Contraindications to study therapies including acute disc herniation, spondylolysis, spondylolithesis, or inflammatory arthritides
* Benign joint hypermobility syndrome

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 185 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
PATIENT-RATED LOW BACK PAIN | 3 and 12 months
  Patients will be asked to rate their typical low back pain over the last week on an 11-box numerical rating scale (0=no pain, 10=the worst pain possible).

SECONDARY OUTCOMES:
Disability | 3 and 12 months
  Disability will be measured with the Roland-Morris- 18 Scale, an 18-item questionnaire that measures the degree to which low back pain restricts patients' daily activities
Quality of Life | 3 and 12 months
  Measured using the 23-item PedsQL instrument which is a developmentally appropriate questionnaire for individuals 8-12 and 13-18 years of age and measures physical, emotional, social and school functioning domains.
Satisfaction with care | 3 and 12 months
  Satisfaction will be measured with a 7-item questionnaire addressing different aspects of patient care including information regarding cause, prognosis, activities, and prevention. Other aspects are concern shown by care provider, quality of recommendations and finally an overall rating of care. Each question will be evaluated on a 5-point Likert scale (1=poor, 5=excellent).
Patient-rated improvement | 3 and 12 months
  Patients will be asked to compare their low back pain condition to what it was before study treatment on a 9-point scale (100% worse to 100% better).
Guardian's satisfaction with care | 3 and 12 months
  Satisfaction will be measured with a 5-item questionnaire addressing concern shown by care provider, quality of recommendations and finally an overall rating of care. Each question will be evaluated on a 5-point Likert scale (1=poor, 5=excellent).
Guardian's impression of Improvement | 3 and 12 months
  Guardians will be asked to compare their child's low back pain condition to what it was before study treatment on a 9-point scale (100% worse to 100% better).
Lumbar Range of Motion | 3 and 6 months
  Lumbar spinal motion will be assessed using the Zebris CMS-HS Spine Motion Analyzer for (1)maximum ranges of motion in the sagittal, coronal, and axial planes and (2) maximum and average velocities and accelerations in the sagittal, coronal, and axial planes from neutral to end-ranges.
Lumbar muscle endurance | 3 and 6 months
  Blinded examiners will measure muscle endurance of the trunk flexors, lateral flexors, and extensors. Specifically, trunk extensors will be measured with the commonly used Biering-Sorensen Test and flexors will be assessed using protocols described by McGill.
Physical activity Level | 3 and 6 months
  Physical activity will be measured by having participants wear a GT1M accelerometer (Actigraph, Inc., Pensacola, FL) for 7 consecutive days. The GT1M is an electronic motion sensor accelerometer.
Expectations | Baseline
  Expectations will be evaluated pre-treatment based on questions that have been used in previous studies by the investigators. Prior to randomization, patients will be asked to rate how helpful they believe each treatment to be on an 11-box scale (0=not at all helpful, 10=extremely helpful). They will also be asked if they had a choice, which treatment would they choose.

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, DC, PhD, Principal Investigator — Northwestern Health Sciences University
Locations (2):
- United States (2):
  - Northwestern Health Sciences University, Bloomington, Minnesota
  - University of Western States, Portland, Oregon

REFERENCES:
- [Derived] Leininger B, Schulz C, Gao Z, Bronfort G, Evans R, Pope Z, Zeng N, Haas M. Accelerometer-Determined Physical Activity and Clinical Low Back Pain Measures in Adolescents With Chronic or Subacute Recurrent Low Back Pain. J Orthop Sports Phys Ther. 2017 Oct;47(10):769-774. doi: 10.2519/jospt.2017.7345. Epub 2017 Sep 12. PMID 28898136
- [Derived] Schulz C, Leininger B, Evans R, Vavrek D, Peterson D, Haas M, Bronfort G. Spinal manipulation and exercise for low back pain in adolescents: study protocol for a randomized controlled trial. Chiropr Man Therap. 2014 May 23;22:21. doi: 10.1186/2045-709X-22-21. eCollection 2014. PMID 24904748